CLINICAL TRIAL: NCT04604288
Title: Individual Patient Expanded Access IND to Evaluate the Safety and Preliminary Efficacy of Autologous HB-adMSCS for the Treatment of Bilateral Knee Pain.
Brief Title: Individual Patient Expanded Access IND of Autologous HB-adMSCS for the Treatment of Bilateral Knee Pain.
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBKP01
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Knee Pain Chronic; Osteo Arthritis Knee
Keywords: Knee; Knee Pain; Osteoarthritis; Stem Cells; MSCs; Intra-articular
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSC — HB-adMSCs (Hope Biosciences autologous adipose-derived mesenchymal stem cells) is manufactured by Hope Biosciences, L.L.C., a biotechnology company headquartered in Sugar Land, Texas.

SUMMARY:
This is an Individual Patient Expanded Access IND of autologous adipose derived Mesenchymal Stem Cells with the primary goal of treating 1 individual with bilateral knee pain who has exhausted all treatment options, his condition has not improved, and his quality of life is severely affected by the condition. There are no FDA approved, fully restorative treatments for his condition. The subject will receive 2 autologous HB-adMSCs intravenous infusion of 200 million (2 x 10^8 cells) total cells, and 4 autologous HB-adMSCs intra-articular injections (1 in each knee joint/ intervention).

DETAILED DESCRIPTION:
* Screening Visit Week 0 The subject will go through a screening process that will last up to 14 days. During this time the Clinical Investigator will review labs and diagnostic test results to confirm study eligibility. Abnormal test results (i.e., ongoing infection), may require follow-up before proceeding with the treatment. This screening period will start with the "Screening Visit", which will include the following procedures:

  1. Informed Consent will be obtained.
  2. Demographics
  3. Review of inclusion and exclusion criteria
  4. Review of medical history and concomitant medications
  5. Physical exam
  6. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
  7. Height and weight
  8. Blood samples will be collected for safety assessments:

     1. Hematology
     2. Chemistry
     3. Coagulation Panel
  9. A verification of patient consent will be verbally performed.
* Intervention 1 Day 1 (Week 1) and Intervention 2 Day 1 (Week 12) Once the eligibility is confirmed, +7 days after the screening visit, the subject will return to

HBSCRF to receive the IV treatment. Procedures will be assessed as follows:

1. Review of medical history, adverse events, and concomitant medications.
2. Physical exam
3. Patient pain assessment VAS of Pain
4. Patient pain assessment WOMAC Knee Score
5. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
6. Weight measurement
7. A verification of patient consent will be verbally performed
8. The HB-adMSCs will be administered and the patient closely observed:

   a. One intravenous infusion of HB-adMSCs (2x108 cells) to last 1 hour:
   1. Volume: 250 ml
   2. Rate: 4-5 mls/min (250ml/h)
9. The subject will then be monitored for a minimum of 1hr after infusion as follows:

   1. Measure Vital signs at minute 0 of the infusion
   2. Measure Vital signs at minute 15 after IV infusion.
   3. Measure Vital Signs at minute 30 after IV infusion.
   4. Measure Vital signs at minute 60 after IV infusion.
   5. Measure Vital signs at minute 120 after IV infusion.
   6. Vital signs will be recorded more frequently if clinically indicated).
10. The Subject will be given comprehensive discharge criteria/instructions.
11. Telephone encounter for adverse events. The subject will be contacted by telephone the following day after the infusion visit to determine if any adverse events have occurred.

    * Post infusion discharge criteria Immediately following the completion of each infusion/injection, the subject should be assessed to ensure that the post-infusion discharge criteria have been met.

    Parameter Values Systolic blood pressure + 20% of baseline. Diastolic blood pressure + 20% of baseline. Heart rate + 20% of baseline Temperature >96.7F and <100.5F Respiratory rate >10 breaths per minute and < 22 breaths per minute Pulse oximetry > 94% on room air

    Additionally, the following will be documented to ensure a safe discharge from the research facility:

    • The patient must be alert and oriented with normal mentation status.
    * The patient must be afebrile with vital signs within normal limits.
    * The patient will be able to ambulate with little or minimal assistance.
    * The patient will rate a level of pain at 3 or below on a scale of 0-10.

      * Intervention 1 Day 2 (Week 1) and Intervention 2 Day 2 (Week 12) 24 hours after the IV infusion the subject will go to the PI's clinic office to receive the intra- articular injections.

        a. Review of medical history, adverse events, and concomitant medications. b. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2) c. Knee MRI without contrast at IA injection 1. If a Knee MRI without contrast has been performed in the last 14 days, it can be used as a baseline and compared with the following Knee MRI without contrast.

        d. The HB-adMSCs will be administered and the patient closely observed:

        a. One ultrasound-guided intra-articular injection in the right knee with 1x108 cells/2ml.

        b. One ultrasound-guided intra-articular injection in the left knee with 1x108 cells/2ml.

        e. The subject will then be monitored for a minimum of 30 minutes after the injections as follows:

        a. Measure Vital signs at minute 0 of infusion. b. Measure Vital signs at minute 15 after IV infusion. c. Measure Vital Signs at minute 30 after IV infusion. d. (Vital signs will be recorded more frequently if clinically indicated). f. The Subject will be given comprehensive discharge criteria/instructions. g. Blood samples will be collected for safety assessments:

        a. Hematology b. Chemistry c. Coagulation Panel h. Telephone encounter for adverse events. i. The subject will be contacted by telephone the following day after the infusion visit to determine if any adverse events have occurred.
        * Post injection discharge criteria Immediately following the completion of each infusion/injection, the subject should be assessed to ensure that the post-infusion discharge criteria have been met.

    Parameter Values Systolic blood pressure + 20% of baseline. Diastolic blood pressure + 20% of baseline. Heart rate + 20% of baseline Temperature >96.7F and <100.5F Respiratory rate >10 breaths per minute and < 22 breaths per minute Pulse oximetry > 94% on room air Additionally, the following will be documented to ensure a safe discharge from the research facility: • The patient must be alert and oriented with normal mentation status. • The patient must be afebrile with vital signs within normal limits.

    • The patient will be able to ambulate with little or minimal assistance.

    • The patient will rate a level of pain at 3 or below on a scale of 0-10.

    -Weeks 3 and 14 - Follow Up Visits

    The patient will be assessed for adverse events 24 hours after each injection with a follow up phone call. The patient will also undergo a thorough on-site follow up visit at the infusion site (HBSCRF) that will include:

<!-- -->

1. Review and update medical history
2. Update concomitant medications list
3. Weight measurement
4. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
5. Physical exam
6. Blood samples will be collected for safety assessments*

   a. Hematology b. Chemistry c. Coagulation Panel
7. Patient pain assessment - Visual Analog Scale
8. WOMAC Knee Score
9. Adverse event monitoring * Safety labs will not be collected at Follow UP Week 14

   -Week 18 - End of the study (EOS)

The patient will undergo an end of study visit at week 18 at the PI's office that will include:

1. Review and update medical history
2. Update concomitant medications list
3. Weight measurement
4. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
5. Physical exam
6. Blood samples will be collected for safety and efficacy assessments:

   1. Hematology
   2. Chemistry
   3. Coagulation Panel
7. Knee MRI without contrast
8. Patient pain assessment - Visual Analog Scale
9. WOMAC Knee Score
10. Adverse Event Monitoring

ELIGIBILITY:
Inclusion Criteria

1. Documented diagnosis of bilateral knee pain.
2. Hemodynamically stable.

Exclusion Criteria

1. Immunosuppression as defined by WBC < 3, 000 cells/ml at baseline screening.
2. Subjects with pro-coagulant disease processes such as Factor V Leiden deficiency, Factor C and S deficiency, anti-thrombin deficiency, prothrombin mutation, and dysfibrinogenemia.
3. Subjects with abnormal vital signs, abnormal liver or kidney function, and hematological abnormalities specifically:

   1. BP systolic: >160 or <100 mmHg, DBP: >100 SBP or <50mmHg
   2. Pulse: <60 or >105 bpm
   3. Respiratory Rate: <9 and >25 breaths per minute
   4. Temperature: >99.9 degrees Fahrenheit
   5. O2 saturation: <92%
   6. Liver enzymes >2x upper limit of normal (ULN)
   7. Abnormal bilirubin unless due to benign unconjugated hyperbilirubinemia
   8. eGFR <60 mL/min/ 1.73 m2 by CKD-EPI
   9. HbA1C >9%
   10. Hb <10 mg/dL
   11. Platelet Count <100,000
4. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation or HB-adMSCs administration.
5. Any abnormal, inexplicable laboratory result with no obvious cause defined.
6. Participation in other interventional research studies.
7. Unwillingness to return for follow-up visits.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Walter R Lowe, MD, Principal Investigator — UT Ortho
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States